CLINICAL TRIAL: NCT04786223
Title: Targeting Neuroinflammation as a Contributing Pathology in Alzheimer's Disease Dementia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Val Lowe (Other)
Responsible Party: Sponsor-Investigator, Val Lowe, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-000866
Record Dates: First submitted 2021-02-18; First posted 2021-03-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Alzheimer's Disease Dementia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- C-11 ER176 PET/CT (Other): C-11 ER176 is an investigational radiopharmaceutical that will be produced under cGMP in the Mayo Clinic Cyclotron Facility. The imaging agent (C-11 ER176) will be administered on an outpatient basis. It will be administered at a single time IV prior to the PET imaging.
  Interventions: Drug: C-11 ER-176; Diagnostic Test: Blood Test

INTERVENTIONS:
Drug: C-11 ER-176 — Participants will receive a one-time administration of C-11 ER176 and undergo a PET/CT imaging study. Blood samples for plasma biomarker testing will be obtained as part of the study.
Diagnostic Test: Blood Test — Participants will undergo a one time venipuncture blood collection to evaluate the presence of inflammatory and genetic markers.

SUMMARY:
This study is being done to research the usefulness of PET/CT imaging for measuring brain inflammation and its relation to Alzheimer's Disease. Additionally, researchers as looking to learn more about the side effects of a new radioactive tracer (radiotracer) C-11 ER176.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) dementia is a devastating illness with no cure. Treatments targeting known pathologic hallmarks of AD, such as amyloid-beta (AB), in symptomatic individuals have proved largely fruitless so other potential disease targets warrant exploration. Neuroinflammation has interesting possible associations with AD dementia and may contribute to AD dementia in different ways among different individuals. Previous PET neuroinflammation data are not entirely consistent and new methods of PET imaging and studies with larger cohorts are needed to further investigate the role of neuroinflammation in AD dementia and the utility of PET as a biomarker. This project seeks to test new PET neuroinflammation imaging methods in unimpaired and AD dementia individuals with biomarker-identified brain pathology to help address these gaps in knowledge in the field.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 60 years of age or older.
* Meet the requirements for one of the four groups (CU A-, CU A+, MCI A+, AD A+).
* Undergoing neurologic evaluation procedures with cognitive testing in the MCSA or - ADRC for a minimum of about 3 years.
* All participants must have had an amyloid PiB PET scan and MRI brain scan within the previous 6 months.
* Capacity to sign consent or have a legally authorized representative to sign the consent.

Exclusion Criteria:

* Participants unable to lie down without moving for 20 minutes.
* Women who are pregnant or cannot stop breast feeding for 24 hours.
* Actively taking daily anti-inflammatory medications (NSAIDs, corticosteroids, etc.) except for a small control group.
* Generalized inflammatory condition and treatment with immunosuppressive, corticoid/glucocorticoid, steroidal or non-steroidal anti-inflammatory medication within 2 weeks of scanning (only acute medication use as an exclusion so as to limit medication interaction but preserve possible chronic systemic inflammation interaction).
* Standard safety exclusionary criteria for MRI such as metallic foreign bodies, pacemaker, etc., since the quantitative PET data analysis is based on anatomic criteria that are established uniquely for each subject by registration to his/her MRI.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Determine if neuroinflammation, as measured by C-11 ER176 SUVr and inflammatory blood test measurements, is correlated with an increase in AB plaque, as measured by C-11 PiB SUVr. | 4 year
  Rationale: Biomarkers that are surrogates of AD pathology are needed to provide methods to select appropriate treatment strategies. We hypothesize that increased neuroinflammation PET signal is seen in AD A+ and MCI A+ as compared to CU A+ participants and is also increased in CU A+ vs. CU A- participants.
Determine if neuroinflammation, as measured by C-11 ER176 SUVr, is correlated with a history of increased cognitive decline in the 5 years preceding PET imaging, as measured by z scores from neuropsychiatric test results (memory, etc.). | 4 year
  Rationale: Surrogate biomarkers of AD pathology, beyond amyloid and tau, are needed to better assess disease progression and prognosis in AD dementia patients. We hypothesize that increased ER176 PET signal in amyloid positive participants is associated with the rate of cognitive decline preceding the neuroinflammation PET scan.
Determine if neuroinflammation, as measured by PET imaging, is associated with plasma biomarkers of inflammation. | 4 year
  Rationale: Plasma biomarkers are advantageous over imaging and CSF biomarkers with regards to cost, invasiveness, and feasibility in community settings. However, they may be less specific. We need to determine how plasma biomarkers correlate with PET neuroinflammation imaging as markers of disease progression, which markers are most highly correlated, and which may be specific to AD pathology. We hypothesize that hsCRP, IL-1B, IL-6, IL-8, IL-10, IL-13, G-CSF, IFN-g, and TNF-a will correlate with increased PET neuroinflammation imaging signal.

SECONDARY OUTCOMES:
Incidence of adverse events attributable to ER176. | 4 year
  Adverse events related to ER176 will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Val Lowe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials